CLINICAL TRIAL: NCT03145116
Title: Clinical Safety and Efficacy of Hydrophilic Acrylic Intraocular Lenses - Retro Prospective Study
Brief Title: Clinical Safety and Efficacy of CT ASPHINA 509 Lenses
Acronym: UVEA509
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment rate
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASPHINA 509-BER-401-17
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 509 (Experimental)
  Interventions: Device: CT ASPHINA 509

INTERVENTIONS:
Device: CT ASPHINA 509 — Intraocular lens

SUMMARY:
Clinical safety and efficacy of CT ASPHINA 509 IOLs after implantation

ELIGIBILITY:
Inclusion Criteria:

Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent;

* Patients of any gender
* Assured follow-up examinations
* Biometry measurement preferably compatible with the IOLMaster evaluation;
* IOL implanted into the capsular bag with IOL model CT ASPHINA 409MP (UVE material) in one eye with at least 12 months follow up at the time of the postop visit
* Patients who had uncomplicated (no peroperative complication) agedrelated cataract surgery in a healthy eye (beside clinically significant cataract)

Exclusion Criteria:

* • BCVA not available preoperatively or better than 0.3 logMAR pre-op

  * Patients unable to meet the limitations of the protocol or likely of noncooperation during the trial
  * Patients whose freedom is impaired by administrative or legal order
  * Concurrent participation in another drug or device investigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 12 to 18 months after surgery
  Monocular best corrected distance visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Augenklinink, Ahaus, Germany

IPD SHARING:
Plan to Share IPD: No